CLINICAL TRIAL: NCT01119664
Title: A Pilot And Feasibility Trial Evaluating Two Different Chemotherapy Regimens In Combination With Intrapleural Adenoviral-Mediated Interferon-Alpha Gene Transfer For Malignant Pleural Mesothelioma
Brief Title: Combination Gene Transfer and Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02510; 811318
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Mesothelioma
Keywords: Adult subjects with malignant pleural mesothelioma who present for first (front) line or second line chemotherapy,
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No prior chemotherapy (Experimental): Intrapleural SCH 721015 (Ad.hIFN-α2b) instilled over 2-5 minutes on Days 1 and 4. Chemotherapy administered for 4 to 6 cycles Subjects with malignant pleural mesothelioma who have been previously untreated with chemotherapy
  Interventions: Drug: SCH 721015
- Patients with prior Pemetrexed-based chemotherapy (Experimental): Intrapleural SCH 721015 (Ad.hIFN-α2b) instilled over 2-5 minutes on Days 1 and 4. Chemotherapy administered for 4 to 6 cycles Subjects with malignant pleural mesothelioma who have been previously treated with chemotherapy
  Interventions: Drug: SCH 721015

INTERVENTIONS:
Drug: SCH 721015

SUMMARY:
The purpose of this study is to find the safety of combination gene therapy and chemotherapy in patients with malignant pleural mesothelioma. Pleural catheter will be placed first, then pts will receive 2 doses of intrapleural vector followed by front line or second line chemotherapy 4-6 cycles every 21 days.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a cancer for which there is no cure. The most effective combination chemotherapy, Pemetrexed (Alimta)/Cisplatin, has yielded overall response rates of up to 40%, but with improvements in overall median survival of only 3.5 months. Prior Phase I trials of intrapleural infusion (IP) of Ad.hIFN-beta (BG00001) were safe. The most recent trial of IP Ad.IFNalpha (SCH 721015) at a dose of 3e11 viral particles (vp) given three days apart was safe and well tolerated, and showed high levels of IFN in pleural fluid and serum. Our preclinical data modeling this proposed study suggest that two IP doses of Ad.IFN-alpha in combination with chemotherapy are well tolerated and markedly enhances efficacy. The purpose of the new study is to determine the safety of administrating intrapleural SCH 721015 (Ad.hIFN-alpha 2b) in combination with chemotherapy for the management of malignant pleural mesothelioma. This study will enroll subjects with pleural mesothelioma. Subjects will receive two fixed dosed of SCH 721015 followed by 4-6 cycles of chemotherapy. Subjects will require placement of a pleural catheter for administration of SCH 721015.

Some patients require a pleural catheter for control of pleural fluid while some will have it placed for research purpose only. Protocol participation is up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* -Pathologically documented malignant mesothelioma
* Must have evaluable disease by RECIST or Modified RECIST Criteria.
* ECOG Performance status equal to or lesser than 1.
* Must be at least 18 years of age.
* Women of childbearing potential and men must use acceptable contraceptive methods during treatment.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial.
* Must be able and willing to give written informed consent.
* No radiotherapy and/or treatment with chemotherapeutic, cytotoxic, or immunologic agents within 4 weeks prior to infusion of the IFN-alpha vector.
* Must have pleural tumor accessible for pleural catheter insertion. Patients with a previously inserted pleural catheter may enroll in the trial and can use the preexisting catheter for vector infusion as long as it is functional and has no evidence of local infection.
* FEV1 equal to or lesser than 1 liter or 40% of predicted value (post-pleural drainage).
* Acceptable hematologic value: granulocyte count equal to or lesser than 1,500/mm3, hemoglobin equal to or lesser than 9 g/dl, platelets equal to or lesser than 100,000/mm3
* Acceptable liver function: bilirubin equal to or less than 1.5 x the upper limit of normal; ALT, AST, and alkaline phosphatase equal to or less than 2.0 x the upper limit of normal
* Acceptable kidney function: creatinine less than 2.0 mg/dl (less than 1.5 mg/dl required for Cisplatin administration) or Creatinine clearance greater than 50.
* Acceptable coagulation status: PT equal to or less than 1.5 x normal, PTT less than 1.5 x normal. However, patients on stable, chronic anti-coagulation therapy with therapeutic anti-coagulation levels will be allowed to enroll in the study.
* Serum albumin must be greater than 2.5 g/dl
* Must have an anti-adenoviral neutralizing antibody titer equal to or less than 1:1000. This will be measured by sub-investigators in the Thoracic Oncology Research Laboratory under standardized (but not GCP) conditions. Results must be known before performing any other research procedures.
* Must have medical insurance coverage (or other means of payment) providing for standard medical interventions in clinical trial, including combination chemotherapy.

Exclusion Criteria:

* Presence of significant pericardial effusion on baseline CT scan of the chest.
* Documented immunodeficiency such as HIV infection.
* Evidence of chronic active Hepatitis B (positive for HBsAg). Prior HBV exposure without evidence of chronic active Hepatitis B is not exclusionary.
* Use of concurrent systemic steroids (greater than10 mg of prednisone per day), immunosuppressives, or any other medications that can directly or indirectly suppress the immune system.
* Presence of any other life-threatening illness, such as unstable angina, severe oxygen dependence, significant chronic obstructive pulmonary disease (COPD), end stage liver or renal disease.
* Rapidly re-accumulating,symptomatic malignant pleural effusion status-post thoracentesis or pleural catheter insertion that requires immediate mechanical or chemical pleurodesis for adequate palliation.
* Presence of untreated brain metastases. Subjects with a prior history of brain metastases will have a CT or MRI scan of the brain to rule out activity.
* Prior bone marrow or stem cell transplants -Female patients who are actively nursing are excluded.
* Patients who have undergone any prior major surgery (excluding pleural catheter placement or infusaport insertion) less than 2 weeks prior to study enrollment.
* Lack of medical insurance coverage (or other form of payment) for standard medical interventions, particularly combination chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2013-10-14 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
To determine the safety of administering intrapleural SCH 721015, Ad.hIFN-alpha2b (Adenoviral-mediated Interferon-alpha) in combination with chemotherapy for the management of MPM. | On going throughout the conduct of the trial
  No dose escalation is planned; however, dose de-escalation is possible should two or more DLTs be encountered in the first six patients treated. With 0 DLTs in 6 patients at a given dose, the upper exact 90% confidence limit on the DLT rate is 32%. With 1 DLT in 6 patients, the Bayesian upper 90% probability limit on the DLT rate is 58%. With 10 subjects per treatment group, we can identify with 90% power any unanticipated toxicity that has prevalence at least 20.6%; with n=15 per group, this figure decreases to 14.2%.

SECONDARY OUTCOMES:
To estimate objective response rates and distribution | On going throughout the conduct of the trial
  Will estimate response rates by 95% confidence intervals, whose half-width will range from as low as 26% (if n=15 subjects are enrolled) to 32% (if n=10).
Time to Progression | On going throughout the conduct of the trial
  Will summarize the distributions of time to progression (TTP) and time to death from any cause by Kaplan-Meier curves. In analyses of TTP, subjects who die without progression will be considered censored at the time of death. Further secondary goals include the evaluation of immunologic indicators of response, including systemic and intrapleural cytokines and cellular and humoral immune responses.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haas, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sterman DH, Alley E, Stevenson JP, Friedberg J, Metzger S, Recio A, Moon EK, Haas AR, Vachani A, Katz SI, Sun J, Heitjan DF, Hwang WT, Litzky L, Yearley JH, Tan KS, Papasavvas E, Kennedy P, Montaner LJ, Cengel KA, Simone CB 2nd, Culligan M, Langer CJ, Albelda SM. Pilot and Feasibility Trial Evaluating Immuno-Gene Therapy of Malignant Mesothelioma Using Intrapleural Delivery of Adenovirus-IFNalpha Combined with Chemotherapy. Clin Cancer Res. 2016 Aug 1;22(15):3791-800. doi: 10.1158/1078-0432.CCR-15-2133. Epub 2016 Mar 11. PMID 26968202